CLINICAL TRIAL: NCT02125032
Title: Transcranial Low Voltage Pulsed Electromagnetic Fields (T-PEMF) in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Bo Mohr Morberg, MD, Ph.D. student, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T-PEMF14; CIV-14-01-011780 (Other: Danish Health and Medicines Authority)
Record Dates: First submitted 2014-04-23; First posted 2014-04-29 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Transcranial pulsed electromagnetic fields (T-PEMF) (Active Comparator): One group receives 8 weeks of active T-PEMF treatment and another group receives 8 weeks of placebo T-PEMF. Both treatments to be performed 30 minutes once a day.
  Interventions: Device: Transcranial low voltage pulsed electromagnetic fields (T-PEMF)
- Trancranial electromagnetic pulsed fields (T-PEMF) (Placebo Comparator): 8 weeks of T-PEMF treatment placebo.
  Interventions: Device: Placebo Transcranial low voltage electromagnetic fields

INTERVENTIONS:
Device: Transcranial low voltage pulsed electromagnetic fields (T-PEMF)
  Other Names: The device name is: Re5 - Parkinson Treatment System
  Arms: Transcranial pulsed electromagnetic fields (T-PEMF)
Device: Placebo Transcranial low voltage electromagnetic fields
  Other Names: The devise name is: Re5 - Parkinson Treatment System
  Arms: Trancranial electromagnetic pulsed fields (T-PEMF)

SUMMARY:
The aim of this study, is to determine whether treatment using transcranial low voltage pulsed electromagnetic fields (T-PEMF) can reduce the symptoms patients with Parkinson's Disease (PD) experience. The symptoms include movement, mentality and the nervous system in general.

Furthermore the purpose of this study is to clarify whether a group of patients with PD, gain a statistical improvement in their symptoms when treated with active T-PEMF, compared to a group of patients with PD who receive placebo T-PEMF .

ELIGIBILITY:
Inclusion Criteria:

* Patients with Idiopathic Parkinson's disease H & Y 1-3 (Hoehn&Yahr)
* MMSE > 22 (a screening test for dementia). (MMSE - Mini-Mental State Examination)
* Age > 18 years.
* The patient is capable understanding, accepting and complete the planned procedures.

Exclusion Criteria:

* The patient has been using T-PEMF before.
* Changes in anti-parkinson drug treatment within the last 6 weeks
* Noticeable dementia or other brain injury, which may affect the ability to give consent, or complicates the assessment of the patient
* Psychosis, or other psychopathological conditions, which requires intervention
* The abuse of alcohol or drugs
* Treatment with Deep Brain stimulation.
* Pregnancy or nursing
* Epilepsy.
* Active implants such as pacemakers and others for example cochlear implants
* Active medical device for example insulin pumps, baclofen pumps.
* Participation in other trials in the intervention period
* Current or previous history of brain tumors, leukemia, malignant melanoma, skin cancer, or head and neck cancer
* Autoimmune disease
* Wounds in the scalp

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2014-05; Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Unified Parkinson´s Disease Rating Scale (UPDRS) | At baseline and at endpoint at week 8.
  Comment on "Title": It is expected that the outcome measure UPDRS will report a change after 8 weeks of treatment compared to baseline.
  Comment on "Time Frame": Data will be assessed at each group after 8 weeks, and will be presented when all included patients have received their intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- OUH Odense University Hospital, Odense C, Funen, Denmark

REFERENCES:
- [Derived] Malling ASB, Morberg BM, Wermuth L, Gredal O, Bech P, Jensen BR. The effect of 8 weeks of treatment with transcranial pulsed electromagnetic fields on hand tremor and inter-hand coherence in persons with Parkinson's disease. J Neuroeng Rehabil. 2019 Jan 31;16(1):19. doi: 10.1186/s12984-019-0491-2. PMID 30704504
- [Derived] Morberg BM, Malling AS, Jensen BR, Gredal O, Bech P, Wermuth L. Effects of transcranial pulsed electromagnetic field stimulation on quality of life in Parkinson's disease. Eur J Neurol. 2018 Jul;25(7):963-e74. doi: 10.1111/ene.13637. Epub 2018 Apr 17. PMID 29573167